CLINICAL TRIAL: NCT01541878
Title: Pilot Study of Breast Cancer Registry in Thailand
Brief Title: Breast Cancer Registry in Thailand
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Prof.Dr. Pornchai O-charoenrat, Professor, Siriraj Hospital
Other Study IDs: ISSARIM0025
Record Dates: First submitted 2012-02-24; First posted 2012-03-01 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Conditions or Focus of Study: *FDAAA; (Enter 1 to 5 Items)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Breast cancer is the most common malignancy affecting women. It is the second leading cause of cancer related death in women in many parts of the world. Breast cancer also occurs in men, accounting for nearly 1% of the total incidence. As a result of continuing research into new treatment methods, women and men with breast cancer now have more treatment options, and a better chance of long-term survival than ever before.

The primary treatment for breast cancer is surgery. Early stage breast cancer, defined for the purposes of this registry as newly diagnosed, clinical stage I to IV breast cancer with no prior therapy for current disease, is often curable with surgery alone. Reports from the National Surgical Adjuvant Breast and Bowel Project (NSABP) and the European Organization for Research and Treatment of Cancer (EORTC) longitudinal trials have explored the efficacy of various surgical techniques as primary treatment of early stage breast cancer1-7. These studies include 20 years of follow-up data that have not shown any significant differences in overall survival or in rates of distant recurrences in women who underwent breast-conserving surgery with radiation therapy versus those who underwent mastectomy. The results of these studies have supported the use of surgery as the standard breast cancer treatment practice around the world.

Data have shown that regardless of the surgical procedure selected for the removal of the primary tumor, micrometastases may be present and lead to the development of disease relapse. In order to decrease the risk of recurrence, patients may receive various therapies. Systemic treatments include chemotherapy and hormonal therapy. Local treatment, such as radiotherapy, can also be used to eliminate malignant cells that remain in the breast, chest wall, or lymph nodes after surgery.

The selection of systemic therapy is a complex process, which is based partly on prognostic factors such as lymph node status, and predictive factors such as hormone receptor status. A number of additional factors are emerging such as HER2/neu overexpression8-10, p53 status, histological evidence of vascular invasion, and quantitative parameters of angiogenesis, but these await confirmation by further research11. However, patient age, socioeconomic status, and availability of treatment options are among a number of other factors that may play a role in determining the type of therapy that a patient is offered.

Over the years, results from a large number of clinical trials have led to the development of various guidelines for breast cancer therapy, including the Early Breast Cancer Trialists Group (EBCTG) conferences in 199512 and 200013, the 2000 National Institutes of Health (NIH) Consensus Conference14, and the 8th St Gallen meeting in 200315. Despite the overview analyses and consensus recommendations, detailed information is lacking regarding the actual use of the currently available breast cancer treatments. Furthermore, the reasons that patients and physicians choose specific therapeutic regimens are not well understood.

With more than 1.2 million people worldwide diagnosed with breast cancer in 200116, and the incidence predicted to increase, making appropriate treatment choices is critical to each breast cancer patient's survival, well-being and quality of life. The plethora of available scientific and lay information can result in a complex and arduous decision-making process for the breast cancer patient and his/her health care provider(s). It is anticipated that this registry will assist in the decision-making process by providing up-to-date information about treatment patterns.

STUDY OBJECTIVES The purpose of the study is to collect, analyze, and disseminate data on patients with stage I-IV breast cancer. The goal of this registry is to improve patients care through a better understanding of treatment patterns and outcomes within individual countries, geographic regions, and ultimately, worldwide.

Primary Objectives:

* Characterize the clinical pattern of patients with breast cancer (clinical stage I-IV as defined by the AJCC17).
* Characterize existing and evolving practice patterns.
* Assess patient disease free and overall survival outcomes.

Secondary Objectives:

* Disseminate findings through publication in peer-reviewed scientific journals.
* Provide supportive data to the development of standard therapies.
* Analyze data and design ancillary studies to address unanswered clinical questions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female > 18 years,
2. Newly diagnosed stage I-IV breast cancer which is defined to meets any one of the following clinical or pathological staging criteria (version 6.0 AJCC classification17) in Appendix B.
3. No prior therapy (other than surgery) for current disease,
4. Written informed consent (if required by local regulations).

Exclusion Criteria:

1. Unable to receive definitive treatment
2. Unable to attend regular follow-up visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with breast cancer undergoing treatment
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-01

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand